CLINICAL TRIAL: NCT01120171
Title: Liposome-encapsulated Doxorubicin (Myocet) Plus Cyclophosphamide as First or Second Line Therapy for Older Patients With Metastatic Breast Cancer
Brief Title: Myocet Plus Endoxan for Older Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.32
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Elderly; Chemotherapy; Cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cyclofosfamide/Liposomal-encapsulated doxorubicin
  Interventions: Drug: Cyclophosphamide; Drug: Liposomal-encapsulated doxorubicin

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide (IV) 600 mg/m2 on day 1. Treatment repeats every 21 days. Primary prophylaxis with pegfilgrastim (6 mg) administered 24 hours after chemotherapy.
  Therapy will continue until maximum response,or unacceptable toxicity.
  Other Names: Endoxan
Drug: Liposomal-encapsulated doxorubicin — Liposomal-encapsulated doxorubicin (IV) 50 mg/m2 on day 1. Treatment repeats every 21 days.
  Primary prophylaxis with pegfilgrastim (6 mg) administered 24 hours after chemotherapy.
  Therapy will continue until maximum response or unacceptable toxicity.
  Other Names: Myocet

SUMMARY:
This study will evaluate the efficacy, safety and effect on quality of life of liposomal-encapsulated doxorubicin in combination with cyclophosphamide as first or second line treatment of older patients (≥ 70 years old) with metastatic breast cancer. The efficacy of the combination will be correlated with the functional status of patients according to the comprehensive geriatric assessment

DETAILED DESCRIPTION:
Elderly individuals make up a large part of the breast cancer population. When treated with chemotherapy for metastatic disease they derive similar benefits to their younger counterparts. Anthracyclines are associated with a cumulative dose-dependent cardiomyopathy with increased rate in patients over the age of 70. Liposomal-encapsulated doxorubicin improves the therapeutic index of doxorubicin by reducing significantly the cardiotoxicity and grade 4 neutropenia and provides comparable antitumor efficacy, when used in combination with cyclophosphamide as first-line therapy for metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic breast adenocarcinoma
* No more than one prior therapy regimen (other than hormonal therapy) for metastatic breast cancer is acceptable.
* Measurable disease as defined by the presence of at least one measurable lesion (except bone metastases, ascites or pleural effusions)
* Performance status (WHO) 0-2
* Adequate liver (serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases)
* Adequate renal function (serum creatinine <1.5 times the upper normal limit)
* Adequate cardiac function (LVEF within normal limits)
* Adequate bone marrow function (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L)
* No radiation of measurable disease (except brain metastases)
* No progressive brain metastases according to clinical or radiological criteria
* No brain metastases without prior radiation therapy
* Written informed consent

Exclusion Criteria:

* Active infection
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* Prior treatment with an anthracycline-containing regimen (as adjuvant therapy) during the previous 12 months period
* Other invasive malignancy except non-melanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI every 3 months

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment every month
Time to Tumor Progression | 1-year
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (11):
- Greece (11):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Heraklion
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Diabalkaniko" hospital, Thessaloniki, Thessaloniki
  - : "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki